CLINICAL TRIAL: NCT00750971
Title: An Open-Label, Phase II Multicenter Cohort Study of Immunoablation With Cyclophosphamide and Antithymocyte-Globulin and Transplantation of Autologous Cd34-Enriched Hemapoietic Stem Cells Versus Currently Available Immunosuppressive/Immunomodulatory Therapy for Treatment of Refractory Systemic Lupus Erythematosus
Brief Title: Autologous Stem Cell Transplantation for Refractory Systemic Lupus Erythematosus (ASSIST)
Acronym: ASSIST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Falk Hiepe, Prof. Dr. Falk Hiepe, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-1306
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: ASSIST; SLE; Stem Cell Transplantation; Tolerance
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Helping Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Immunoablation and Autologous Hematopoietic Stem Cell Transplantation
  Interventions: Procedure: Immunoablation and Autologous Hematopoietic Stem Cell Transplantation
- 2 (Active Comparator): Best currently available immunosuppressive/immunomodulatory therapy
  Interventions: Procedure: Immunoablation and Autologous Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Immunoablation and Autologous Hematopoietic Stem Cell Transplantation — Transplantation of purified CD34+ autologous hematopoietic stem cells mobilized with cyclophosphamide (200mg/m2)and G-CSF (10µg/kg/d) after immunoablation with cyclophosphamide (200mg/kg)and rabbit-antithymocyteglobulin (90mg/kg)

SUMMARY:
While glucocorticoids and immunosuppressants ameliorate manifestations of SLE in many patients, current therapies are insufficient to control the disease in a subset of patients, and their clinical prognosis remains poor due to the development of vital organ failure, cumulative drug toxicity and to the increased risk of cardiovascular disease and malignancy. Immunoablative chemotherapy followed by autologous hematopoietic stem cell transplantation (ASCT) has recently emerged as a promising experimental therapy for severely affected patients, providing them the potential to achieve treatment-free, long-term remission. The investigators postulate that immunoablative therapy eliminates or effectively reduces the level of autoreactive T and B lymphocytes and then regeneration of de novo immunity resets the autoreactive immune system into a self-tolerant, protective immune system resulting in prolonged and treatment-free remission.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SLE according to American College of Rheumatology (ACR) classification criteria
2. Age between 18 and 60 years, inclusive
3. Provision of informed consent
4. Active disease, refractory to standard immunosuppressive therapy defined as:

   * BILAG level A and a SLEDAI-score of at least 10, despite treatment with high-dose corticosteroids and pulse intravenous CYC at doses of 500-1000mg/m2 for at least 6 months or mycophenolate mofetil (MMF) at doses of at least 2g -
   * Lupus nephritis with renal biopsy performed within one year prior to screening showing glomerulonephritis WHO class III or IV
   * Parenchymal disease of heart or lung
   * Neuropsychiatric lupus
   * Autoimmune cytopenia OR
   * recurrence of disease activity (defined as BILAG level A and a SLEDAI of at least 10) within one year after successful induction therapy with cyclophosphamide or MMF in the presence of an adequate maintenance therapy with either cyclophosphamide (at least 500mg/m2 monthly), mycophenolate mofetil (at least 2g daily), azathioprine (at least 1.5mg/kg/d), methotrexate (at least 15mg weekly), cyclosporine (at least 3mg/kg/d) in patients with persistent anti-dsDNA antibodies

Exclusion Criteria:

1. Severe concomitant disease or organ damage

   * renal: renal insufficiency with glomerular filtration rate below 40ml/min
   * cardiac: congestive heart failure, LVEF < 40% determined by echocardiogram, uncontrolled arrhythmia
   * pulmonary: mean pulmonary arterial pressure >50mmHg, DLCO < 40 % predicted
   * gastrointestinal: liver cirrhosis; SGOT, SGPT greater than 2 x the upper limit of normal, unless due to active lupus
2. Ongoing cancer or history of malignancy within 5 years of screening
3. Women who are pregnant or breastfeeding or use non-reliable methods of contraception
4. Subjects with active systemic infection
5. Subjects with history of active viral infection within 6 months prior to screening, known HIV-infection or chronic Hepatitis B or Hepatitis C
6. History of allergic reaction to cyclophosphamide, G-CSF or ATG
7. Use of immunosuppressive agents for indications other than SLE
8. Any comorbidity that in the opinion of the investigator would jeopardize the ability of the subject to tolerate therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
SLEDAI | 48 months

SECONDARY OUTCOMES:
Serologic response (autoantibodies) | 48 months
Immune Reconstitution | 48 months
Organ-specific response parameters | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Falk Hiepe, Prof, Principal Investigator — Universitätsmedizin Charité
Locations (8):
- Germany (8):
  - Universitätsmedizin Charité, Berlin
  - Universitätsklinik Köln, Cologne
  - Universitätsklinik Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinik Heidelberg, Heidelberg
  - Universitäsklinik Mainz, Mainz
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinik Würzburg, Würzburg

REFERENCES:
- [Background] Thiel A, Alexander T, Schmidt CA, Przybylski GK, Kimmig S, Kohler S, Radtke H, Gromnica-Ihle E, Massenkeil G, Radbruch A, Arnold R, Hiepe F. Direct assessment of thymic reactivation after autologous stem cell transplantation. Acta Haematol. 2008;119(1):22-7. doi: 10.1159/000117824. Epub 2008 Feb 22. PMID 18292651
- [Background] Jayne D, Passweg J, Marmont A, Farge D, Zhao X, Arnold R, Hiepe F, Lisukov I, Musso M, Ou-Yang J, Marsh J, Wulffraat N, Besalduch J, Bingham SJ, Emery P, Brune M, Fassas A, Faulkner L, Ferster A, Fiehn C, Fouillard L, Geromin A, Greinix H, Rabusin M, Saccardi R, Schneider P, Zintl F, Gratwohl A, Tyndall A; European Group for Blood and Marrow Transplantation; European League Against Rheumatism Registry. Autologous stem cell transplantation for systemic lupus erythematosus. Lupus. 2004;13(3):168-76. doi: 10.1191/0961203304lu525oa. PMID 15119545
- [Background] Rosen O, Thiel A, Massenkeil G, Hiepe F, Haupl T, Radtke H, Burmester GR, Gromnica-Ihle E, Radbruch A, Arnold R. Autologous stem-cell transplantation in refractory autoimmune diseases after in vivo immunoablation and ex vivo depletion of mononuclear cells. Arthritis Res. 2000;2(4):327-36. doi: 10.1186/ar107. Epub 2000 Jun 8. PMID 11056673
- [Background] Alexander T, Thiel A, Rosen O, Massenkeil G, Sattler A, Kohler S, Mei H, Radtke H, Gromnica-Ihle E, Burmester GR, Arnold R, Radbruch A, Hiepe F. Depletion of autoreactive immunologic memory followed by autologous hematopoietic stem cell transplantation in patients with refractory SLE induces long-term remission through de novo generation of a juvenile and tolerant immune system. Blood. 2009 Jan 1;113(1):214-23. doi: 10.1182/blood-2008-07-168286. Epub 2008 Sep 29. PMID 18824594